CLINICAL TRIAL: NCT06574295
Title: Health Technology Assessment of Pulmonary Nodules Using Non-intubated Video-assisted Thoracic Surgery Based on the Real-world Evidence
Brief Title: HTA of NIVATS Based on RWE
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yingyao Chen, Professor, Fudan University
Other Study IDs: FudanU-2024-07-1145
Record Dates: First submitted 2024-08-26; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Pulmonary nodule; VATs
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-intubated Video-assisted Thoracic Surgery Group: This group will undergo non-intubated video-assisted thoracic surgery (VATS), a minimally invasive procedure that avoids the use of endotracheal intubation and mechanical ventilation. Instead, patients maintain spontaneous breathing throughout the surgery under regional anesthesia or sedation. The technique is designed to reduce anesthesia-related complications, improve recovery times, and enhance overall patient comfort compared to traditional intubated thoracic surgeries.
- Intubated Thoracic Surgery Group: This group will undergo traditional intubated thoracic surgery, where patients are intubated and placed on mechanical ventilation under general anesthesia. This method is commonly used in thoracic surgeries to control the airway and ensure adequate ventilation during the procedure. However, it may be associated with a higher incidence of anesthesia-related complications, such as airway trauma and slower postoperative recovery, compared to non-intubated techniques.

SUMMARY:
This research focuses on a Health Technology Assessment (HTA) of non-intubated video-assisted thoracic surgery (VATS) for lung nodules. Lung cancer, one of the most prevalent malignancies globally, has a high incidence and mortality rate, particularly in China. Traditional treatments like thoracotomy are highly invasive, while conventional thoracoscopic surgery can induce anesthesia-related complications. Non-intubated VATS offers a promising alternative by avoiding intubation and mechanical ventilation, thus reducing complications, anesthesia burden, and recovery time.

The study aims to comprehensively assess the clinical effectiveness, safety, and economic viability of non-intubated VATS for lung cancer treatment through systematic literature reviews, real-world evidence (RWE), and cost-effectiveness analysis. The research will also explore patient preferences using discrete choice experiments (DCE).

By evaluating this technology from a Chinese perspective, the study seeks to provide evidence-based recommendations for the broader adoption of non-intubated VATS in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

- Experimental Group (Non-intubated Video-assisted Thoracic Surgery)：

1. Patients diagnosed with pulmonary nodules or lung cancer who are scheduled for minimally invasive surgery (including wedge resection, segmentectomy, or lobectomy).
2. Aged between 18 and 75 years, regardless of gender.
3. Preoperative assessment indicates that the patient can tolerate non-intubated video-assisted thoracic surgery.
4. The patient has signed an informed consent form and voluntarily agrees to participate in the study.

Control Group (Intubated Video-assisted Thoracic Surgery)：

1. Patients diagnosed with pulmonary nodules or lung cancer who are scheduled for minimally invasive surgery (including wedge resection, segmentectomy, or lobectomy).
2. Aged between 18 and 75 years, regardless of gender.
3. Preoperative assessment indicates that the patient can tolerate minimally invasive surgery.
4. The patient has signed an informed consent form and voluntarily agrees to participate in the study.

Exclusion Criteria:

1. Patients unable to provide sufficient preoperative and postoperative follow-up data.
2. Pregnant or breastfeeding women.
3. Patients with severe cardiopulmonary dysfunction preoperatively, making them unfit for surgery.
4. Patients who have previously undergone surgery or radiotherapy in the same chest region.
5. Patients with active infections or other severe comorbidities that may affect surgical outcomes.
6. Patients with mental illness or cognitive impairment who cannot understand the study content or comply with follow-up requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 75 years who have been diagnosed with pulmonary nodules or lung cancer and are scheduled for minimally invasive thoracic surgery. These patients will be divided into two groups: an experimental group undergoing non-intubated video-assisted thoracic surgery (VATS) and a control group undergoing intubated VATS. Both groups include individuals who are able to tolerate surgery based on preoperative evaluations, regardless of gender. All participants must provide informed consent and agree to complete the required follow-up assessments.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
Patient-reported Outcomes | Measured within 3 days post-surgery
  The primary outcome will be assessed using two validated instruments: the Anderson Symptom Inventory (lung cancer-specific module) and the EQ-5D. The Anderson Symptom Inventory will measure symptom severity (e.g., pain, fatigue, nausea, sleep disturbance) and the impact of symptoms on daily functioning, while the EQ-5D will evaluate overall health-related quality of life, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The scores will provide insight into patients' recovery and well-being following non-intubated video-assisted thoracic surgery (VATS) compared to traditional intubated thoracic surgery.
Postoperative hospitalization time | Measured in days from surgery completion to hospital discharge.
  The secondary outcome will measure the duration of the postoperative hospital stay. This will be assessed as the number of days from the completion of surgery to the patient's discharge. The goal is to compare the efficiency of recovery between patients undergoing non-intubated video-assisted thoracic surgery (VATS) and those receiving traditional intubated thoracic surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Yingyao Chen, PhD, Study Chair — School of Public Health，Fudan University
Locations (1):
- School of Public Health, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No